CLINICAL TRIAL: NCT00900263
Title: S0120, A Prospective Observational Biologic Study of Asymptomatic Patients With Monoclonal Gammopathy and Plasmaproliferative Disorders
Brief Title: S0120, Studying Blood and Bone Marrow Samples From Patients With Monoclonal Gammopathy of Undetermined Significance, Multiple Myeloma, or Plasmacytoma
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S0120; S0120 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma; Plasma Cell Myeloma; Precancerous Condition
Keywords: stage I multiple myeloma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance
MeSH Terms: conditions — Multiple Myeloma; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance | interventions — Cytogenetic Analysis; Microarray Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow/peripheral blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: microarray analysis
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow in the laboratory from patients with monoclonal gammopathy of undetermined significance, multiple myeloma, or plasmacytoma may help doctors learn more about changes that occur in DNA and identify biomarkers related to these diseases. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at blood and bone marrow samples from patients with monoclonal gammopathy of undetermined significance, multiple myeloma, or plasmacytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish a serum, cell, and bone marrow tissue bank of prospectively collected samples from patients with monoclonal gammopathy of undetermined significance (MGUS), asymptomatic multiple myeloma, solitary plasmacytoma, or other plasma cell dyscrasias.
* Evaluate the feasibility of accruing patients with these diseases.
* Determine whether patterns of gene expression or cytogenetics exist that allow molecular delineation of MGUS subtypes.
* Characterize cellular and humoral immune response to known tumor antigens in these patients.
* Cryopreserve serum/T cells for future evaluation.
* Preliminarily identify biological correlates that may relate to progression to symptomatic disease.

OUTLINE: Patients are stratified according to diagnosis (monoclonal gammopathy of undetermined significance [MGUS] or other plasma cell dyscrasias vs asymptomatic multiple myeloma vs solitary plasmacytoma).

Blood and bone marrow samples are collected and analyzed for microarray analysis, cytogenetic analysis, and immunobiology studies.

Unused samples may be stored for future research studies.

Patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following plasmaproliferative diseases:

  * Monoclonal gammopathy of undetermined significance (MGUS)
  * Asymptomatic multiple myeloma
  * Solitary plasmacytoma
  * Other plasma cell dyscrasias
* Disease does not require therapy
* Willing to submit research samples for gene expression analysis and immunologic assessment

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other malignancy within the past 2 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or adequately treated stage I or II cancer from which the patient is currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for this disease

Chemotherapy

* No prior chemotherapy for this disease

Endocrine therapy

* No prior endocrine therapy for this disease

Radiotherapy

* No prior radiotherapy for this disease

Surgery

* No prior surgery for this disease

Other

* Prior or concurrent bisphosphonates allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: plasmaproliferative disease not requiring therapy
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2002-06; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Disease progression | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Dhodapkar, MD, Study Chair — Rockefeller University
Locations (69):
- United States (69):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Highlands Oncology Group - Springdale, Bentonville, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Clemens Regional Medical Center, Mount Clemens, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Background] Spisek R, Kukreja A, Chen LC, Matthews P, Mazumder A, Vesole D, Jagannath S, Zebroski HA, Simpson AJ, Ritter G, Durie B, Crowley J, Shaughnessy JD Jr, Scanlan MJ, Gure AO, Barlogie B, Dhodapkar MV. Frequent and specific immunity to the embryonal stem cell-associated antigen SOX2 in patients with monoclonal gammopathy. J Exp Med. 2007 Apr 16;204(4):831-40. doi: 10.1084/jem.20062387. Epub 2007 Mar 26. PMID 17389240
- [Background] Zhan F, Barlogie B, Arzoumanian V, Huang Y, Williams DR, Hollmig K, Pineda-Roman M, Tricot G, van Rhee F, Zangari M, Dhodapkar M, Shaughnessy JD Jr. Gene-expression signature of benign monoclonal gammopathy evident in multiple myeloma is linked to good prognosis. Blood. 2007 Feb 15;109(4):1692-700. doi: 10.1182/blood-2006-07-037077. Epub 2006 Oct 5. PMID 17023574
- [Derived] Dhodapkar MV, Sexton R, Hoering A, Van Rhee F, Barlogie B, Orlowski R. Race-Dependent Differences in Risk, Genomics, and Epstein-Barr Virus Exposure in Monoclonal Gammopathies: Results of SWOG S0120. Clin Cancer Res. 2020 Nov 15;26(22):5814-5819. doi: 10.1158/1078-0432.CCR-20-2119. Epub 2020 Aug 18. PMID 32816893
- [Derived] Dhodapkar MV, Sexton R, Das R, Dhodapkar KM, Zhang L, Sundaram R, Soni S, Crowley JJ, Orlowski RZ, Barlogie B. Prospective analysis of antigen-specific immunity, stem-cell antigens, and immune checkpoints in monoclonal gammopathy. Blood. 2015 Nov 26;126(22):2475-8. doi: 10.1182/blood-2015-03-632919. Epub 2015 Oct 14. PMID 26468228
- [Derived] Dhodapkar MV, Sexton R, Waheed S, Usmani S, Papanikolaou X, Nair B, Petty N, Shaughnessy JD Jr, Hoering A, Crowley J, Orlowski RZ, Barlogie B. Clinical, genomic, and imaging predictors of myeloma progression from asymptomatic monoclonal gammopathies (SWOG S0120). Blood. 2014 Jan 2;123(1):78-85. doi: 10.1182/blood-2013-07-515239. Epub 2013 Oct 21. PMID 24144643